CLINICAL TRIAL: NCT02737722
Title: A Phase I/IIa, Randomized Double Blind, Placebo-Controlled, Dose Escalating Study to Evaluate the Safety and Tolerability of Topically Applied Bisphosphocin Nu-3 on Infected Diabetic Ulcers of Subjects With Type I or II Diabetes Mellitus
Brief Title: Topically Applied Bisphosphocin Nu-3 on Infected Diabetic Ulcers of Subjects With Type I or II Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lakewood-Amedex Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAI2014-1
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-10

CONDITIONS: Diabetic Foot Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bisphosphocin Nu-3 (Experimental): Dosage Form: Topical Antimicrobial, Dosage: 1mg/mL, 10 mg/mL, 20 mg/mL, 50 mg/mL, 100 mg/mL Frequency: QD for day 1, 2x daily for 7 days, Duration: 8 days
  Interventions: Drug: Bisphosphocin Nu-3
- Placebo (Placebo Comparator): Dosage Form: Diluent, Frequency: QD for day 1, 2x daily for 7 days, Duration: 8 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bisphosphocin Nu-3
  Other Names: Nu-3
  Arms: Bisphosphocin Nu-3
Drug: Placebo
  Arms: Placebo

SUMMARY:
Phase I/IIa, five cohort ascending dose with two dosing arms per cohort, study in Type I or II diabetes mellitus subjects with a chronic infected diabetic ulcer defined as having a DUSS score of 0 to 3 and DFI wound score of 1 to 3.

DETAILED DESCRIPTION:
The study is designed to run the cohorts in series with the completion of the first cohort before initiating the next dosing level. At all study visits the ulcer will be visually examined for any changes and photographed using the Aranz Medical Silhouette™ system that will calculate area and depth of the ulcer.

In Arm 1, eligible subjects will be treated with a single application of Nu-3 or placebo in 4 to 1 ratio to judge the initial safety of Nu-3 over a brief one (1) hour interval and 24-hr interval post application. Bisphosphocin Nu-3 will be applied topically to the chronic infected ulcer, covered with a non-abrasive bandage following the initial observation period. The subject will be released with verbal instructions to leave the bandage on the wound and return for a follow up visit within 24h ± 2h. At the follow up visit, the bandage will be removed, the ulcer visually examined and the subject cleared for the MAD Arm 2 based on the recommendation of the PI and absence of any SAEs.

In Arm 2, eligible subjects which are those who have been approved by the PI after the Visit 2 examination will be instructed in the proper application of bisphosphocin Nu-3. The subjects will be observed applying the first dose in the clinic to ensure compliance. Subjects will then be given a 7 day supply and sent home to continue treatment. Visit 4 or earlier in the case of any adverse events, subjects will return to the clinic for an examination, including visual examination of the ulcer, vital signs, adverse events, photo documentation, collection of a sample for microbiology and concomitant medication use. A final follow up visit will be scheduled +7 days after last dose of study medication (Day 15) for a complete examination as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 85.
2. Voluntary written consent, given before performance of any clinical investigation-related procedure not part of standard medical care, and with the understanding that consent may be withdrawn at any time without prejudice to future medical care.
3. Non-hospitalized ambulatory subjects suffering from Diabetes mellitus, Type I or II
4. Diabetic foot ulcer(s) with a DUSS Score of 0 to 3
5. Ulcerated area(s) of not more than two (2) ulcers between 0.5 to 6 cm2
6. Any female of child bearing age must consent to use medically acceptable birth control for the duration of the study
7. Female subjects must meet at least one of the following additional criteria:

   1. Surgically sterile with bilateral tubal ligation or hysterectomy.
   2. Post-menopausal for at least one year.
   3. If of child-bearing potential, practicing an acceptable method of birth control for the duration of the clinical investigation as judged by the Investigator, such as condoms, foams, jellies, diaphragm, intrauterine device or abstinence.
8. Subjects willing to undergo pre-and post-clinical investigation blood collection, physical exams and laboratory investigations.

Exclusion Criteria:

1. A DUSS Score above 3.
2. DUSS Probing to Bone = "Yes"
3. An ulcer area(s) greater than 6 cm2 or more than two (2) ulcers
4. Any subject that has received systemic or topical antibiotics within the last seven (7) days
5. Any subject on topical antimicrobial treatment for their infected diabetic foot ulcer whose ulcer is responding to treatment
6. Any subject that would be unable to follow the protocol procedures, safely monitor the infection status at home, and return for schedule visits
7. Positive pregnancy test at Screening or Visit 2
8. Active infection as demonstrated by temperature > 37.5 oC and clinical features of active infection.
9. Known immunosuppression or taking immunosuppressive agents including systemic steroids.
10. History of severe co-morbidity with expected patient survival ≤ 6 months.
11. Pregnancy or lactation
12. Intake of investigational drugs within 28 days prior to enrollment.
13. History of concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol.
14. Likely inability to comply with the protocol or cooperate fully with the investigator and site personnel.
15. Unwillingness or language barrier precluding adequate understanding of the trial procedure or cooperation with trial site personnel.
16. Known or suspected active abuse of alcohol, narcotics or non-prescription drugs.
17. Other planned surgical procedures within 30 days prior to or 30 days post-index procedure.
18. Prior enrollment in this clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Kates, PhD, Study Director — Lakewood-Amedex Inc
Locations (3):
- United States (3):
  - Center for Clinical Research, Inc., San Francisco, California
  - Journey Research, Inc., Oldsmar, Florida
  - Clinical Research Solutions, Franklin, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 48 participants were screened; 17 were screen failures and weren't enrolled. One participant was enrolled but not randomized.
Groups:
- 0.1% Bisphosphocin Nu-3: Participants received a single topical administration of 0.1% Nu-3 solution in saline on Day 1. Participants then applied the same dose twice a day for 7 days.
- 1% Bisphosphocin Nu-3: Participants received a single topical administration of 1% Nu-3 solution in saline on Day 1. Participants then applied the same dose twice a day for 7 days.
- 2% Bisphosphocin Nu-3: Participants received a single topical administration of 2% Nu-3 solution in saline on Day 1. Participants then applied the same dose twice a day for 7 days.
- Placebo: Participants received a single topical administration of matching placebo on Day 1. Participants then applied the same dose twice a day for 7 days.
Period: Overall Study
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo
Started | 8 | 8 | 8 | 6
Completed | 8 | 8 | 7 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (8.21) | 59.3 (8.41) | 60.5 (14.03) | 61.0 (6.54) | 59.0 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 0 | 6
  Male | 7 | 5 | 6 | 6 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 0 | 7 | 7 | 3 | 17
  Unknown or Missing | 8 | 0 | 0 | 3 | 11
Mean Diabetic Ulcer Wound Scoring System (DUSS) Score [Mean (Standard Deviation); unit: units on a scale] — Ulcers were scored based on the DUSS. The following 4 parameters were scored as either 0 or 1. Palpable pedal pulses: presence, 0; absence, 1. Probing to the bone: no, 0; yes, 1. Location of ulcer: toe, 0; foot, 1. Number of ulcerations: single, 0; multiple, 1. The four parameter scores were summed to calculate a total score ranging from 0 to 4, with a higher score indicating increased severity. Baseline is defined as the last non-missing value obtained prior to receiving study drug. Data are collected in the Intent-to-Treat Population, comprised of all randomized participants.
  units on a scale | 1.13 (0.35) | 1.25 (0.71) | 1.13 (0.64) | 1.00 (0.89) | 1.13 (0.63)
Mean Diabetic Foot Ulcer Wound Infection Score [Mean (Standard Deviation); unit: units on a scale] — Baseline is defined as the last non-missing value obtained prior to receiving study drug. The score for each parameter is summed to calculate a total score, from 0 (less severe infection) to 19 (more severe infection). Parameters: purulent discharge (0, absent; 3, present); non-purulent discharge (serious, sanguineous) (0, absent; 1, mild); other signs/symptoms of inflammation (erythema, induration, tenderness, pain; 0, none; 1, mild; 2, moderate; 3, severe); local warmth (relative to uninfected contralateral foot) (0, same; 1, mildly increased; 2, moderately increased; 3, severely increased).
  units on a scale | 4.38 (0.92) | 4.50 (1.60) | 4.63 (1.69) | 4.33 (1.31) | 4.47 (1.31)
Mean Ulcer Area in the Intent-to-Treat Population [Mean (Standard Deviation); unit: centimeters squared (cm^2)] — Baseline is defined as the last non-missing value obtained prior to receiving study drug.
  centimeters squared (cm^2) | 1.5 (1.23) | 1.8 (1.54) | 1.9 (1.25) | 0.8 (0.20) | 1.5 (1.22)
Mean Ulcer Area in the Per-Protocol Population [Mean (Standard Deviation); unit: cm^2] — Population: Data were collected in the Per-Protocol Population, comprised of all participants who met enrollment criteria, received all doses of investigational product as required by the protocol, and had no major protocol violations.
  cm^2
    number analyzed (Participants) | 5 | 8 | 8 | 6 | 27
    (all) | 1.7 (1.36) | 1.8 (1.54) | 1.9 (1.25) | 0.8 (0.20) | 1.6 (1.24)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Treatment-emergent Adverse Events as Graded According to the Common Terminology Criteria for Adverse Events v4.02 (CTCAE)
Description: The severity of each adverse event, as judged by the investigator, was graded according to the CTCAE v4.02. Treatment-emergent adverse events are defined as adverse events with onset times after dosing, or pre-existing adverse events that worsened during the study.
Time Frame: up to Day 15 (Visit 5)
Population: Safety Population: all participants administered any amount of investigational product
Measure: Count of Participants; unit: Participants
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Normal and Abnormal Cultures at Visits 2, 3, 4, and 5
Description: The microbiological response to bisphosphocin Nu-3 based on aerobic and anaerobic culture and sensitivity was determined by measuring the reduction of pathogenic bacteria following Nu-3 treatment. Each laboratory used their own standards to decide whether the cultures were normal or abnormal.
Time Frame: Days 1, 2, 9, and 15 (Visits 2, 3, 4, and 5, respectively)
Population: Intent-to-Treat (ITT) Population: all randomized participants. Only those participants with available data were analyzed. Microbiology results were not collected in the database for participants in the 0.1% cohort.
Measure: Number; unit: participants
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo
Number analyzed (Participants) | 0 | 8 | 8 | 6
participants
  Day 1 (Visit 2), Normal Culture: number analyzed (Participants) | 0 | 8 | 7 | 4
  Day 1 (Visit 2), Normal Culture |  | 2 | 0 | 0
  Day 1 (Visit 2), Abnormal Culture: number analyzed (Participants) | 0 | 8 | 7 | 4
  Day 1 (Visit 2), Abnormal Culture |  | 6 | 7 | 4
  Day 2 (Visit 3), Normal Culture: number analyzed (Participants) | 0 | 8 | 8 | 4
  Day 2 (Visit 3), Normal Culture |  | 1 | 2 | 1
  Day 2 (Visit 3), Abnormal Culture: number analyzed (Participants) | 0 | 8 | 8 | 4
  Day 2 (Visit 3), Abnormal Culture |  | 7 | 6 | 3
  Day 9 (Visit 4), Normal Culture: number analyzed (Participants) | 0 | 8 | 7 | 2
  Day 9 (Visit 4), Normal Culture |  | 1 | 0 | 0
  Day 9 (Visit 4), Abnormal Culture: number analyzed (Participants) | 0 | 8 | 7 | 2
  Day 9 (Visit 4), Abnormal Culture |  | 7 | 7 | 2
  Day 15 (Visit 5), Normal Culture: number analyzed (Participants) | 0 | 7 | 7 | 4
  Day 15 (Visit 5), Normal Culture |  | 1 | 0 | 1
  Day 15 (Visit 5), Abnormal Culture: number analyzed (Participants) | 0 | 7 | 7 | 4
  Day 15 (Visit 5), Abnormal Culture |  | 6 | 7 | 3
Statistical Analysis 1: Comparison: 1% Bisphosphocin Nu-3 vs Placebo; Day 1 (Visit 2); Test type: Superiority; p = 0.5152, Fisher Exact
Statistical Analysis 2: Comparison: 2% Bisphosphocin Nu-3 vs Placebo; Day 1 (Visit 2); Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: 1% Bisphosphocin Nu-3 vs Placebo; Day 2 (Visit 3); Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 4: Comparison: 2% Bisphosphocin Nu-3 vs Placebo; Day 2 (Visit 3); Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 5: Comparison: 1% Bisphosphocin Nu-3 vs Placebo; Day 9 (Visit 4); Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 6: Comparison: 2% Bisphosphocin Nu-3 vs Placebo; Day 9 (Visit 4); Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 7: Comparison: 1% Bisphosphocin Nu-3 vs Placebo; Day 15 (Visit 5); Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 8: Comparison: 2% Bisphosphocin Nu-3 vs Placebo; Day 15 (Visit 5); Test type: Superiority; p = 0.3636, Fisher Exact

3. Secondary Outcome: Mean Change From Baseline in the Diabetic Ulcer Severity Score (DUSS)
Description: Clinical response to bisphosphocin Nu-3 was determined by visual evaluation of ulcers, based on the Principal Investigator's judgement, following Nu-3 treatment. Ulcers were scored based on the DUSS. The following 4 parameters were scored as either 0 or 1. Palpable pedal pulses: presence, 0; absence, 1. Probing to the bone: no, 0; yes, 1. Location of ulcer: toe, 0; foot, 1. Number of ulcerations: single, 0; multiple, 1. The four parameter scores were summed to calculate a total score ranging from 0 to 4, with a higher score indicating increased severity. Baseline is defined as the last non-missing value obtained prior to receiving study drug. Change from Baseline is calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Day 15 (Visit 5)
Population: ITT Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo
Number analyzed (Participants) | 8 | 8 | 7 | 6
score on a scale | 0.13 (0.64) | -0.13 (0.35) | -0.14 (0.69) | -0.33 (0.52)
Statistical Analysis 1: Comparison: 0.1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.172, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: 1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.365, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: 2% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.619, Wilcoxon Rank Sum Test

4. Secondary Outcome: Mean Change From Baseline in the Diabetic Foot Ulcer Wound Infection Score
Description: Change from Baseline is calculated as the post-Baseline value minus the Baseline value. Baseline is defined as the last non-missing value obtained prior to receiving study drug. The Diabetic Foot Ulcer Wound Infection Score is a numerical scoring system comprised of 7 wound parameters. The score for each individual parameter is summed to calculate a total score, ranging from 0 (less severe infection) to 19 (more severe infection). Parameters are as follows: purulent discharge (0, absent; 3, present); non-purulent discharge (serious, sanguineous) (0, absent; 1, mild); other signs and symptoms of inflammation (erythema, induration, tenderness, pain; 0, none; 1, mild; 2, moderate; 3, severe); local warmth (relative to uninfected contralateral foot) (0, same; 1, mildly increased; 2, moderately increased; 3, severely increased).
Time Frame: Baseline; Day 15 (Visit 5)
Population: ITT Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo
Number analyzed (Participants) | 8 | 8 | 7 | 6
score on a scale | -2.38 (1.41) | -1.50 (3.42) | -2.86 (1.57) | -3.00 (2.10)
Statistical Analysis 1: Comparison: 0.1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.432, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: 1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.435, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: 2% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.715, Wilcoxon Rank Sum Test

5. Secondary Outcome: Mean Change From Baseline in Ulcer Area in the ITT Population
Description: Change from Baseline is calculated as the post-Baseline value minus the Baseline value. Baseline is defined as the last non-missing value obtained prior to receiving study drug. For participants who have more than one ulcer, the measurement of all ulcers were combined for analysis.
Time Frame: Baseline; Day 15 (Visit 5)
Population: ITT Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: centimeters squared (cm^2)
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo
Number analyzed (Participants) | 8 | 8 | 7 | 6
centimeters squared (cm^2) | -0.3 (0.62) | -0.2 (0.77) | -0.7 (0.68) | -0.3 (0.32)
Statistical Analysis 1: Comparison: 0.1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.519, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: 1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.519, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: 2% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.153, Wilcoxon Rank Sum Test

6. Secondary Outcome: Mean Change From Baseline in the Percentage of Area Reduction for Ulcers in the ITT Population
Description: as for outcome 5
Time Frame: Baseline; Day 15 (Visit 5)
Population: ITT Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of area
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo
Number analyzed (Participants) | 8 | 8 | 7 | 5
percentage of area | 25.2 (34.41) | 10.8 (51.94) | 54.0 (36.67) | 41.0 (41.56)
Statistical Analysis 1: Comparison: 0.1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.464, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: 1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.464, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: 2% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.465, Wilcoxon Rank Sum Test

7. Secondary Outcome: Mean Change From Baseline in Ulcer Area in the Per-Protocol Population
Description: as for outcome 5
Time Frame: Baseline; Day 15 (Visit 5)
Population: Per-Protocol Population: all participants who met enrollment criteria, received all doses of investigational product as required by the protocol, and had no major protocol violations. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: centimeters squared (cm^2)
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo
Number analyzed (Participants) | 5 | 8 | 7 | 6
centimeters squared (cm^2) | -0.1 (0.37) | -0.2 (0.77) | -0.7 (0.68) | -0.3 (0.32)
Statistical Analysis 1: Comparison: 0.1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.361, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: 1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.519, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: 2% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.153, Wilcoxon Rank Sum Test

8. Secondary Outcome: Mean Change From Baseline in the Percentage of Area Reduction for Ulcers in the Per-Protocol Population
Description: as for outcome 5
Time Frame: Baseline; Day 15 (Visit 5)
Population: Per-Protocol Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of area
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo
Number analyzed (Participants) | 5 | 8 | 7 | 5
percentage of area | 22.4 (39.77) | 10.8 (51.94) | 54.0 (36.67) | 41.0 (41.56)
Statistical Analysis 1: Comparison: 0.1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.465, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: 1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.464, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: 2% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.465, Wilcoxon Rank Sum Test

9. Post Hoc Outcome: Percentage of Participants With a Positive and Negative Global Clinical Impression of Microbiology Response
Description: Global impression of microbiological response was conducted by comparing culture value from Baseline to Visit 5 (Day 15). If culture values were not reported by the local laboratory, numerical values were assigned using the following criteria: heavy growth, 4+, moderate growth, 2+, scant, 1+, no bacteria, 0.
Time Frame: Baseline; Day 15 (Visit 5)
Population: Per-Protocol Population. Microbiology results were not collected in the database for participants in the 0.1% cohort.
Measure: Number; unit: percentage of participants
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo
Number analyzed (Participants) | 0 | 8 | 8 | 6
percentage of participants
  No apparent effect (negative) |  | 62 | 38 | 75
  Apparent effect (positive) |  | 38 | 62 | 25

10. Post Hoc Outcome: Median Percent Change From Baseline in the Percentage Area Reduction for Ulcers in the Per-Protocol Population
Description: Percent change from Baseline is calculated as the [(post-Baseline value minus the Baseline value)/Baseline value] x 100. Baseline is defined as the last non-missing value obtained prior to receiving study drug. For participants who have more than one ulcer, the measurement of all ulcers were combined for analysis.
Time Frame: Baseline; Day 15 (Visit 5)
Population: Per-Protocol Population. Only those participants with available data were analyzed.
Measure: Median (Full Range); unit: percent change
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo
Number analyzed (Participants) | 5 | 8 | 7 | 5
percent change | 4.6 [-13.5 to 87.9] | 13.1 [-77.2 to 89.2] | 65.6 [-4.0 to 90.1] | 29.9 [-10.8 to 84.5]
Statistical Analysis 1: Comparison: 0.1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.465, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: 1% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.464, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: 2% Bisphosphocin Nu-3 vs Placebo; Test type: Superiority; p = 0.465, Wilcoxon Rank Sum Test

ADVERSE EVENTS:
Time Frame: up to Day 15 (Visit 5)
Description: Treatment-emergent adverse events, defined as adverse events with onset times after dosing, or pre-existing adverse events that worsened during the study, are reported.
Arm/Group | 0.1% Bisphosphocin Nu-3 | 1% Bisphosphocin Nu-3 | 2% Bisphosphocin Nu-3 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/8 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.1% Bisphosphocin Nu-3 (N=8) | 1% Bisphosphocin Nu-3 (N=8) | 2% Bisphosphocin Nu-3 (N=8) | Placebo (N=6)
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.1% Bisphosphocin Nu-3 (N=8) | 1% Bisphosphocin Nu-3 (N=8) | 2% Bisphosphocin Nu-3 (N=8) | Placebo (N=6)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Participants were enrolled into Cohorts 1, 2, and 3; Cohorts 4 and 5 were not enrolled because of challenges with enrolling participants. Additionally, Lakewood Amedex developed a gel formulation to be used for subsequent clinical studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT02737722/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT02737722/SAP_001.pdf